CLINICAL TRIAL: NCT06570746
Title: "Comparison of the Effectiveness of Conventional Radiofrequency Thermocoagulation and Chemical Ablation With Phenol on Articular Branches of Femoral and Obturator Nerves in Chronic Hip Pain"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Akylai Dosieva, doctor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
Keywords: Radiofrequency thermocoagulation; Phenol chemical ablation
MeSH Terms: conditions — Chronic Pain | interventions — Hypnotics and Sedatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency thermocoagulation to the articular branches of the femoral and obturatory nerves (Experimental): Patients are operated under sedation in the operating room. C-arm fluoroscopy device is used for imaging purposes for radiofrequency thermocoagulation process. In order to prevent vascular injury the needle is advanced under the guidance of ultrasonography. There are target points determined in fluoroscopy for the femoral nerve and the obturatory nerve. Before the thermocoagulation procedure, local anesthetic and steroid are injected into each of the target points.
  Interventions: Drug: Sedative
- Chemical ablation with phenol (Active Comparator): Patients are operated under sedation in the operating room. C-arm fluoroscopy device is used for imaging purposes for radiofrequency thermocoagulation process. In order to prevent vascular injury the needle is advanced under the guidance of ultrasonography. There are target points determined in fluoroscopy for the femoral nerve and the obturatory nerve. Before the thermocoagulation procedure, local anesthetic and steroid are injected into each of the target points. Before the procedure, the femoral artery was visualized with a linear ultrasound probe to prevent arterial injury by entering 2 cm lateral to the femoral artery. Following this, a mixture of 2.5 cc of 0.05% bupivacaine and 2.5 cc of 6% phenol was applied, and a lesion was created for 90 seconds at 80°.
  Interventions: Drug: Sedative

INTERVENTIONS:
Drug: Sedative — Sedation is applied before the procedure

SUMMARY:
"In our study, we aimed to compare the effects of conventional radiofrequency thermocoagulation applied to the articular branches of the femoral and obturator nerves with chemical ablation using phenol on hip pain."

DETAILED DESCRIPTION:
"Our study is designed as a double-blind, prospective randomized controlled trial. Blinding will be ensured by keeping the researcher performing pain diary follow-ups unaware of which procedure was applied to each patient.

Patients will be randomized using computer-assisted methods. Following approval from the hospital ethics committee, clinical trial registration will be conducted. From 2024 to 2025, patients presenting with chronic hip pain to the Department of Algology at ADU Faculty of Medicine will be divided into two groups. In Group 1, chemical ablation of the femoral and obturator nerve branches with phenol under ultrasound guidance will be performed. In Group 2, conventional radiofrequency thermocoagulation of the articular branches of the femoral and obturator nerves under ultrasound guidance will be applied.

During the study, pain intensity will be assessed using the Numerical Rating Scale (NRS) at baseline, 2 hours post-procedure, and at 1 month and 3 months post-procedure for both Group 1 and Group 2. The WOMAC scale will be used to evaluate their functional capacity."

ELIGIBILITY:
Inclusion Criteria:

Be older than 18 years old. Written consent must be obtained. Have had chronic hip pain for more than 3 weeks. -

Exclusion Criteria:

Major psychiatric illness Presence of lumbar radicular pain or referred pain in the patient Patients using anticoagulant agents Patients with infection in the area where the procedure will be performed Those with allergy to local anesthetics Those allergic to phenol or betamethasone Pregnant women Scheduled for surgery

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
NRS (Numerical Rating Scale) | preoperative
  We will assess NRS (Numerical Rating Scale) scores at 1 month and 3 months. A 50% reduction in NRS will be considered statistically significant
NRS (Numerical Rating Scale) | postoperative first month
  We will assess NRS (Numerical Rating Scale) scores at 1 month and 3 months. A 50% reduction in NRS will be considered statistically significant
NRS (Numerical Rating Scale) | postoperative third month
  We will assess NRS (Numerical Rating Scale) scores at 1 month and 3 months. A 50% reduction in NRS will be considered statistically significant

SECONDARY OUTCOMES:
WOMAC (Western OntarioandMcMasterUniversitiesArthritis Index ) | preoperative
  To assess functional capacity preoperatively, we will evaluate the WOMAC (Western Ontario and McMaster Universities Arthritis Index) scale at 1 month and 3 months post-procedure in patients.
WOMAC (Western OntarioandMcMasterUniversitiesArthritis Index ) | postoperative first month
  To assess functional capacity preoperatively, we will evaluate the WOMAC (Western Ontario and McMaster Universities Arthritis Index) scale at 1 month and 3 months post-procedure in patients.
WOMAC (Western OntarioandMcMasterUniversitiesArthritis Index ) | postoperative third month
  To assess functional capacity preoperatively, we will evaluate the WOMAC (Western Ontario and McMaster Universities Arthritis Index) scale at 1 month and 3 months post-procedure in patients.

CONTACTS AND LOCATIONS:
Overall Officials: akylai dosieva, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Faculty of Medicine, Aydin, Turkey (Türkiye)